CLINICAL TRIAL: NCT01520233
Title: Genome Based Outcome Prediction in High Risk Neuroblastoma
Brief Title: Gene Expression in Predicting Outcome in Samples From Patients With High-Risk Neuroblastoma
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: ANBL12B2; COG-ANBL12B2 (Other: Children's Oncology Group); CDR0000723895 (Other: Clinical Trials.gov); ANBL12B2 (Other: Children's Oncology Group); NCI-2012-00240 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-01-26; First posted 2012-01-27 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Neuroblastoma
Keywords: disseminated neuroblastoma; localized unresectable neuroblastoma; recurrent neuroblastoma; regional neuroblastoma; stage 4S neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — Gene Expression Profiling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: RNA analysis
Genetic: gene expression analysis
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of tumor tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in RNA and predict how patients will respond to treatment. It may also help doctors find better ways to treat cancer.

PURPOSE: This research trial studies gene expression in predicting outcomes in samples from patients with high-risk neuroblastoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* To test the correlation of a previously published microarray gene expression signature with the gene expression obtained with the nCounter™ Analysis System using RNA isolated from formalin-fixed, paraffin-embedded (FFPE), high-risk neuroblastoma samples.
* To construct, test, and validate a novel robust classifier that can be readily integrated into the clinic.

OUTLINE: This is a multicenter study.

RNA samples extracted from paraffin-embedded tissue are analyzed for gene signature expression levels by nCounter™ Analysis System and correlated with published microarray expression data. Results are then used to develop a refined gene-expression-profile classifier of ultra high-risk neuroblastoma.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Formalin-fixed paraffin-embedded tumor sections linked to clinical and outcome data collected from high-risk neuroblastoma patients (n=100) treated at the University of Chicago, St. Jude Children's Research Hospital, Children's Memorial Hospital, or Texas Children's Hospital

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Neuroblastoma patients treated at the University of Chicago, St. Jude Children's Research Hospital, Children's Memorial Hospital, or Texas Children's Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2012-01; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Linear correlation between the nCounter™ Analysis System and the expression data obtained in microarray platforms
nCounter™ Analysis System and microarray platforms equally predictive of outcome in the high-risk group of neuroblastoma patients

CONTACTS AND LOCATIONS:
Overall Officials: Susan L. Cohn, MD, Principal Investigator — University of Chicago Comer Children's Hospital